CLINICAL TRIAL: NCT02562443
Title: A Phase III, International, Randomized, Controlled Study of Rigosertib Versus Physician's Choice of Treatment in Patients With Myelodysplastic Syndrome After Failure of a Hypomethylating Agent
Brief Title: Controlled Study of Rigosertib Versus Physician's Choice of Treatment in MDS Patients After Failure of an HMA
Acronym: INSPIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Top line analysis indicated that the study had failed to achieve its primary endpoint.
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-30; 2015-001476-22 (EudraCT Number)
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Myelodysplastic Syndrome; MDS; Refractory Anemia With Excess Blasts; RAEB
Keywords: Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rigosertib + best supportive care (BSC) (Experimental)
  Interventions: Drug: rigosertib; Drug: best supportive care (BSC)
- Physician's Choice (PC) + best supportive care (BSC) (Active Comparator)
  Interventions: Drug: Any approved or standard-of-care therapy; Drug: best supportive care (BSC)

INTERVENTIONS:
Drug: rigosertib — Patients will receive intravenous rigosertib 1800 mg/24 hr for 3 days every 2 weeks for first 8 cycles, then every 4 weeks thereafter + best supportive care (BSC).
  Other Names: ON 01910.Na
  Arms: rigosertib + best supportive care (BSC)
Drug: Any approved or standard-of-care therapy — Patients will receive Physician's Choice of Treatment or alternative treatment which may include any approved or standard-of-care therapy, based on frequently used treatment for MDS (no experimental therapy) + best supportive care.
  Arms: Physician's Choice (PC) + best supportive care (BSC)
Drug: best supportive care (BSC) — Patients will receive best supportive care (BSC): azacitidine (AZA) and/or decitabine (DAC) are permitted.
  Arms: Physician's Choice (PC) + best supportive care (BSC)
Drug: best supportive care (BSC) — Patients will receive best supportive care (BSC).
  Arms: rigosertib + best supportive care (BSC)

SUMMARY:
The study's primary objective [in a population of patients with MDS after failure of treatment with azacitidine (AZA) or decitabine (DAC)], is to compare the overall survival (OS) of patients in the rigosertib group vs the Physician's Choice group, in all patients and in a subgroup of patients with IPSS-R very high risk.

DETAILED DESCRIPTION:
This is a Phase III, open-label, randomized, controlled, international study. Approximately 360 patients < 82 years of age with MDS classified as RAEB-1, RAEB-2, or RAEB-t who received AZA or DAC for ≤ 9 months and/or ≤ 9 cycles over 12 months and had their last dose of AZA or DAC within 6 months prior to screening will be stratified by:

* Very high risk (VHR) vs non-VHR per IPSS-R, and
* Geographic region (North America vs Europe vs Asia; because approved products and standard of care may vary by region), and randomly assigned in a 2:1 ratio to one of the following 2 treatment groups:
* Rigosertib 1800 mg/24 hr administered as a 72 hr CIV infusion on Days 1, 2, and 3 of a 2 week cycle for the first 8 cycles, and on Days 1, 2, and 3 of a 4-week cycle thereafter (N = approximately 240 patients);
* Physician's Choice of alternative treatment, which may include any approved or standard-of-care therapy that the patient has not shown to be hypersensitive to, based on frequently used treatment for MDS, as per institutional guidelines, after receipt of HMAs (N = approximately 120 patients). The drugs used in the Physician's Choice arm should be used according to the recommendations, if clinically appropriate, provided in the corresponding Summary of Product Characteristics (SmPC) and Prescribing Information of these drugs. Experimental therapies are not allowed on the PC arm.

Patients will be treated until 2006 IWG progression criteria are met (ie, 50% increase of BM blasts or worsening of cytopenias) or until an unacceptable toxicity or intolerance.

For all randomized patients who discontinue study treatment, subsequent therapies with their start and end dates, as well as survival time after treatment discontinuation, will be documented at least monthly until death.

Patients in the PC group who progress will not be allowed to cross over to rigosertib.

All patients in both treatment groups will be allowed, as medically justified, access to RBC and platelet transfusions and to growth factors (granulocyte colony-stimulating factor (G-CSF), erythropoietin, and thrombopoietin).

ELIGIBILITY:
Inclusion Criteria:

* MDS classified as follows:

  * RAEB-1 per World Health Organization (WHO) MDS criteria (5% to <10% BM blasts)
  * RAEB-2 per WHO MDS criteria (10% to <20% BM blasts)
  * RAEB-t per French-American-British (FAB) classification (20% to 30% BM blasts)
* At least one cytopenia (ANC < 1800/µL or platelet count < 100,000/µL or hemoglobin [Hgb] < 10 g/dL)
* Progression (according to 2006 IWG criteria) at any time after initiation of AZA or DAC treatment or Failure to achieve complete or partial response or hematological improvement (HI) (according to 2006 IWG) after at least six 4-week cycles of AZA or either four 4-week or four 6-week cycles of DAC administered or Relapse after initial complete or partial response or HI (according to 2006 IWG criteria)
* Duration of prior HMA therapy ≤ 9 months and/or total ≤ 9 cycles of prior HMA therapy in ≤ 12 months
* Last dose of AZA or DAC within 6 months before the planned date of randomization; however, must be off these treatments for ≥ 4 weeks before randomization
* Has failed to respond to, relapsed following, not eligible for, or opted not to participate in allogeneic stem cell transplantation
* Off all treatments for MDS (including AZA and DAC) for ≥ 4 weeks before randomization; growth factors (G-CSF, erythropoietin and thrombopoietin) and transfusions are allowed before and during the study as clinically indicated
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Willing to adhere to protocol prohibitions and restrictions
* Patient must sign informed consent form to indicate patient's understanding study's purpose and procedures and willingness to participate. Should patient be incapable of giving consent, the patient's legally authorized representative (as defined by local regulation) must give consent. However, should patient, in any manner, choose not to participate this takes precedence and will be respected.
* Patients with 5q- syndrome should have failed to respond to or progressed on treatment with lenalidomide, where available and indicated

Exclusion Criteria:

* Previous participation in a clinical study of IV or oral rigosertib; patients who failed screening for other rigosertib studies may be screened for participation
* Eligible to receive induction chemotherapy, such as 7-10 days of cytosine arabinoside plus 2-3 days of an anthracycline, or high-dose cytarabine
* Suitable candidate to receive allogeneic stem cell transplantation; patient is eligible for study if a suitable candidate refuses to undergo an allogeneic stem cell transplant or a suitable donor cannot be found
* Any active malignancy within the past year, except basal cell or squamous cell skin cancer or carcinoma in situ that is unlikely to progress in two years
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure or unstable angina pectoris
* Active infection not adequately responding to appropriate therapy
* Total bilirubin ≥1.5 mg/dL not related to hemolysis or Gilbert's disease
* Alanine transaminase (ALT)/aspartate transaminase (AST) ≥2.5 x upper limit of normal (ULN)
* Serum creatinine ≥2.0 mg/dL or eGFR (estimated Glomerular Filtration Rate) < 40 mL/min.
* Known active HIV, hepatitis B or hepatitis C, where active is defined as follows:

  * HIV or hepatitis C - presence of viral load
  * Hepatitis B - antigen positive
* Uncorrected hyponatremia (defined as serum sodium value of <130 mEq/L)
* Female patients of child-bearing potential and male patients with sexual partners of child-bearing potential who are unwilling to follow strict contraception requirements before entry and throughout the study, up to and including the 30-day non-treatment follow-up period. Examples of acceptable contraception methods include:

  * estrogen-gestagen based contraceptives associated with inhibition of ovulation (oral, intravaginal, transdermal),
  * gestagen-only based contraceptives associated with inhibition of ovulation (oral, injectable, implantable),
  * intra-uterine devices (IUDs),
  * intra-uterine hormone-releasing systems (IUSs),
  * bilateral tubal occlusion
  * vasectomized partner
  * sexual abstinence in accordance with an individual's lifestyle
* Female patients of child-bearing potential (pre-menopausal and not surgically sterilized) who are breast-feeding or have a positive blood beta-human chorionic gonadotropin pregnancy test at Screening
* Major surgery without full recovery or within 3 weeks before planned randomization;
* Uncontrolled hypertension
* New onset seizures (within 3 months before planned randomization) or poorly controlled seizures
* Any other concurrent investigational agent or chemotherapy, radiotherapy, immunotherapy, or corticosteroids (prednisone up to 20 mg/day or its equivalent is permitted for chronic conditions)
* Treatment with cytarabine at any dose, lenalidomide, or any other therapy targeted to the treatment of MDS (other than growth factors and other supportive care measures) within 4 weeks of planned randomization
* Investigational therapy within 4 weeks of planned randomization
* Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements.
* Patient previously diagnosed with AML (defined as a bone marrow or peripheral blood blast percentage of >30%).

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Overall survival of all randomized patients and overall survival of patients scored as IPSS-R very high risk. | Up to 30 Months
  The overall survival (OS) of all randomized patients (ITT population), and the overall survival of patients scored as IPSS-R very high risk.

SECONDARY OUTCOMES:
Overall survival of patients with monosomy 7 chromosomal aberrations. | Up to 30 Months
  Evaluate OS of patients with monosomy 7 chromosomal aberrations in the rigosertib vs PC group. Overall survival is the time (months) from date of randomization to date of death or date last known to be alive at the time of date cut-off.
Overall survival of patients with trisomy 8 chromosomal aberrations. | Up to 30 Months
  Evaluate OS of patients with trisomy 8 chromosomal aberrations in the rigosertib vs PC group. Overall survival is the time (months) from date of randomization to date of death or date last known to be alive at the time of date cut-off.
Percent of patients with response according to 2006 IWG criteria. | Up to 30 Months
  Responses of complete remission (CR), partial remission (PR), mCR, SD, failure, and PD will be determined by 2006 IWG criteria. The number and percent of patients with CR, PR, mCR, SD, Failure, or PD will be summarized by treatment group.
Scores of Quality of Life Questionnaire. | At Baseline, at Week 4, Every 4 Weeks thereafter, and at the End-of-treatment.
  Compare rigosertib vs PC in regard to the the scores of the EuroQol EQ-5D-5L Questionnaire. The EuroQol EQ-5D-5L Questionnaire includes five levels of severity in each of the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and a visual analogue scale.
Percent of patients with bone marrow blast response rate according to 2006 IWG criteria. | Up to 30 Months
  Compare rigosertib vs PC in regard to the bone marrow blast responses of marrow complete response (mCR ≥ 50% decrease of BMBL vs pretreatment values to a value ≤ 5%), marrow partial response (mPR, ≥ 50% decrease of BMBL vs pretreatment values to a value > 5%), stable disease (SD, no mCR or mPR, but no progressive disease (PD), and PD (≥ 50% BMBL increase relative to baseline or nadir) will be assessed. The number and percent of patients with mCR, mPR, SD, or PD will be summarized by treatment group. Responses of complete remission (CR), partial remission (PR), mCR, SD, failure, and PD will be determined by 2006 International Working Group (IWG) criteria.
Percent of patients with hematologic improvement (HI) (erythroid, platelet and neutrophil responses) according to 2006 IWG criteria. | Up to 30 Months
  Compare rigosertib vs PC in regard to the number and percent of patients who meet the 2006 IWG criteria.

OTHER OUTCOMES:
Exploratory Objective: Bone Marrow Genomic Mutational Status | At screening, every 8 week during study treatment, and at the end of study treatment
  Bone marrow genomic mutational status.
Exploratory Objective: Transition to Acute Myelogenous Leukemia (AML) | Through study completion, an average of 8 months
  Transformation time to AML (defined as a bone marrow or peripheral blood blast percentage >30%).
Safety Objective: Number of Patients with AEs. | Monthly, through study completion
  Treatment-emergent adverse events (TEAEs) will be graded according to NCI CTCAE version 4, grouped by MedDRA preferred term, and summarized by worst grade of severity per patient by treatment group.
Safety Objective: Rigosertib population pharmacokinetics (PK). | At Cycle 1 (Week 1) and Cycle 2 (Week 3), on Day 1 of the infusion, 1 hr after its start and on Day 2 of the infusion, 6 hr after its start
  Blood samples for population PK analysis will be taken in rigosertib patients

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Fruchtman, MD, Study Chair — Traws Pharma, Inc.
Locations (158):
- United States (32):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - Mid Florida Hematology and Oncology Centers, Orange City, Florida
  - Advanced Research Institute, Inc, St. Petersburg, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Loyola University Chicago at Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health Hospital, Indianapolis, Indiana
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota Physicians Bone Marrow Transplant Clinic, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Cancer Center, Philadelphia, Pennsylvania
  - Greenville Health System (GHS) Cancer Institute, Greenville, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Seattle Cancer Care Alliance (SCCA), Seattle, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Australia (3):
  - Icon Cancer Care Icon South Brisbane, South Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Health, Monash Medical Centre, Melbourne, Victoria
- Austria (3):
  - Hospital of the Elisabethinen Linz GmbH, Linz
  - Salzburg University Hospital, Salzburg
  - Hanusch Hospital, Vienna
- Belgium (4):
  - Antwerp Hospital Network Stuivenberg, Antwerp
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Campus Gasthuisberg, Leuven
  - CHU UCL Namur - Site Godinne, Yvoir
- Canada (4):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Croatia (4):
  - Klinički bolnički centar Osijek, Osijek
  - Clinical Hospital Merkur, Zagreb
  - Klinički bolnicki centar Sestre milosrdnice, Zagreb
  - Klinički bolnički centar Zagreb, Zagreb
- Czechia (5):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Ostrava, Department of Hematooncology, Ostrava Poruba
  - General University Hospital, Prague
  - Institute of Hematology and Blood Transfusion, Prague
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Tartu University Hospital, Tartu
- France (9):
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital Claude Huriez, CHRU Lille, Lille
  - Institut Paoli-Calmettes, Marseille
  - Hôpital l'Archet 1, Nice
  - Institut de Cancérologie du Gard, Nîmes
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Hôpital civil, Strasbourg, Strasbourg
  - CHRU Tours Hôspital Bretonneau, Tours
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Marien Hospital Düsseldorf, Düsseldorf
  - Universitätsklinikum Frankfurt am Main, Frankfurt
- Hungary (4):
  - Semmelweis University Medical School, Budapest
  - Somogy County Kaposi Mór Teaching Hospital, Kaposvár
  - Jósa András Teaching Hospital, Nyíregyháza
  - University of Pécs 1st Department of Internal Medicine, Pécs
- India (7):
  - Hemato Oncology Clinic Pvt. Ltd, Ahmedabad, Gujarat
  - St. John's Medical College Hospital, Bangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Jaslok Hospital and Research Center, Mumbai, Maharashtra
  - Sahyadri Clinical Research and Development Center, Pune, Maharashtra
  - Christian Medical College, Vellore, Tamil Nadu
  - Institute Of Hematology And Transfusion Medicine, Kolkata, West Bengal
- Ireland (3):
  - Cork University Hospital, Cork
  - Adelaide and Meath Hospital, Incorporating the National Children's Hospital, Dublin
  - University Hospital Waterford, Waterford
- Israel (7):
  - Ha'Emek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (9):
  - Polyclinic S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili, Brescia
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara
  - A.O.U. Pisana, Divisione di Ematologia - University Hospital of Pisa, Pisa
  - Policlinico Universitario Tor Vergata, Roma
  - Ospedale S. Eugenio - S. Eugenio Hospital, Roma
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Cittá della Salute e della Scienza di Torino, Torino
- Japan (31):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Chugoku Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuyama, Hiroshima
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Shimane University Hospital, Izumo, Shimane
  - Japanese Red Cross Medical Center, Shibuya City, Tokyo
  - Akita University Hospital, Akita
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō City
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - Tokai Central Hospital of the Mutual Aid Association of Public School Teachers, Kakamigahara
  - Saitama Medical Center, Kawagoe
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Niigata University Medical and Dental Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - Kindai University Hospital, Osakasayama-shi
  - Oita Prefectural Hospital, Ōita
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - NTT Medical Center Tokyo, Shinagawa-ku
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Dokkyo Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - Yamagata University Hospital, Yamagata
  - Saiseikai Yokohamashi Nanbu Hospital, Yokohama
  - University of Fukui Hospital, Yoshida
- Poland (5):
  - Independent Public Healthcare Facility University Hospital in Cracow, Clinical Department of Hematology, Krakow
  - Independent Public Health Care Facility of the Ministry of Internal Affairs with Warmia and Mazury Oncology Centre in Olsztyn, Olsztyn
  - Ludwik Rydygier Provinicial Hospital in Suwalki, Department of Clinical Oncology and Hematology, Suwałki
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Independent Public University Hospital No. 1 in Wroclaw, Department of Hematology, Blood Cancers and Bone Marrow, Wroclaw
- Russia (3):
  - State Autonomous Healthcare Institution of Kemerovo region "Kemerovo Regional Clinical Hospital n.a. S.V. Belyaev",, Kemerovo
  - State Budgetary Healthcare Institution of Moscow City, Moscow
  - FSBI "Russian Scientific Research Hematology and Tranfusiology Institute of the Federal Biomedical Agency", Saint Petersburg
- Spain (9):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Duran i Reynals - Instituto Catalán de Oncología, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitari i Politècnic La Fe, Valencia
- Sweden (4):
  - Karolinska University Hospital, Stockholm, Huddinge
  - Skåne University Hospital, Department of Hematology, Lund
  - Uppsala University Hospital, Uppsala
  - Linköping University Hospital, Linköping, Östergötland County
- Switzerland (2):
  - University Hospital and University of Bern; Inselspital Bern, Bern
  - University Hospital Zurich, Zurich
- United Kingdom (5):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - The Royal Liverpool University Hospital, Liverpool
  - St Bartholomew's Hospital, Barts Health NHS Trust, London
  - King's College Hospital NHS Foundation Trust, London

REFERENCES:
- [Background] Garcia-Manero G, Fenaux P, Al-Kali A, Baer MR, Sekeres MA, Roboz GJ, Gaidano G, Scott BL, Greenberg P, Platzbecker U, Steensma DP, Kambhampati S, Kreuzer KA, Godley LA, Atallah E, Collins R Jr, Kantarjian H, Jabbour E, Wilhelm FE, Azarnia N, Silverman LR; ONTIME study investigators. Rigosertib versus best supportive care for patients with high-risk myelodysplastic syndromes after failure of hypomethylating drugs (ONTIME): a randomised, controlled, phase 3 trial. Lancet Oncol. 2016 Apr;17(4):496-508. doi: 10.1016/S1470-2045(16)00009-7. Epub 2016 Mar 9. PMID 26968357
- [Background] Athuluri-Divakar SK, Vasquez-Del Carpio R, Dutta K, Baker SJ, Cosenza SC, Basu I, Gupta YK, Reddy MV, Ueno L, Hart JR, Vogt PK, Mulholland D, Guha C, Aggarwal AK, Reddy EP. A Small Molecule RAS-Mimetic Disrupts RAS Association with Effector Proteins to Block Signaling. Cell. 2016 Apr 21;165(3):643-55. doi: 10.1016/j.cell.2016.03.045. PMID 27104980
- [Background] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.